CLINICAL TRIAL: NCT03114878
Title: The Value of Eye Movement Desensitization Reprocessing in the Treatment of Tinnitus
Brief Title: The Value of EMDR in the Treatment of Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Tine Luyten, Tine Luyten Clinical Psychologist, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECUZA16/35/360
Record Dates: First submitted 2016-12-20; First posted 2017-04-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Eye Movement Desensitization Reprocessing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- TRT / EMDR (Active Comparator): Tinnitus Retraining Therapy / Eye Movement Desensitization Reprocessing
  Interventions: Behavioral: TRT / CBT
- TRT / CBT (Active Comparator): Tinnitus Retraining Therapy / Cognitive Behavioral Therapy
  Interventions: Other: TRT / EMDR

INTERVENTIONS:
Other: TRT / EMDR — Tinnitus Retraining Therapy:
  TRT is a therapy developed by Prof. Pawel Jastrebroff and Dr. Jonathan Hazell. During the counseling, the patient is educated about the work mechanism of tinnitus and how to deal with the emotional and physical responses. The main goal is to habituate to the sound of the ringing in the ears.
  Eye Movement Desensitization and Reprocessing:
  This is a scientifically, psychotherapeutic approach, developed in 1987 by Francine Shapiro. EMDR represents a specific method within a wider theoretical model called 'Adaptive Information Processing (AIP)'. Within the treatment bilateral stimulation is used i.e. visual, auditory and tactile stimuli can be used to stimulate both the left - and the right hemisphere.
  Other Names: TRT / Eye Movement Desensitization Reprocessing
  Arms: TRT / CBT
Behavioral: TRT / CBT — Tinnitus Retraining Therapy:
  TRT is a therapy developed by Prof. Pawel Jastrebroff and Dr. Jonathan Hazell. During the counseling, the patient is educated about the work mechanism of tinnitus and how to deal with the emotional and physical responses. The main goal is to habituate to the sound of the ringing in the ears.
  Cognitive Behavioral Therapy:
  CBT is the combination of behavioral therapy with interventions that have been developed from cognitive psychology. The founders of CBT are Aaron Beck and Albert Ellis. The core idea is the assumption that so-called negative cognitions are responsible for dysfunctional behavior. The techniques used in the cognitive behavioral therapy focus on changing the content of these irrational cognitions.
  Other Names: TRT / Cognitive Behavioral Therapy
  Arms: TRT / EMDR

SUMMARY:
A prospective, randomized, controlled, clinical trial with blind evaluator that uses TRT and EMDR as a treatment for tinnitus.

DETAILED DESCRIPTION:
Patients with subjective, chronic, non-pulsatile tinnitus will be randomized in two treatment groups: TRT and CBT versus TRT and EMDR. Evaluations will take place at baseline before therapy starts, at the end of the treatment, after 3 months (10 treatment sessions) and 3 months after therapy ends. The Tinnitus Functional Index (TFI) will be used as the primary outcome measurement. Secondary outcome measurements will be the Visual Analogue Scale of Loudness (VAS), Tinnitus Questionnaire (TQ), Hospital Anxiety and Depression Scale (HADS), Hyperacusis Questionnaire (HQ), psychoacoustic measurements and Event-related potentials (ERP). The objective is to evaluate whether the bimodal therapy TRT and EMDR can provide faster and/or more relief from the annoyance experienced in chronic tinnitus patients' daily lives compared to the bimodal therapy TRT and CBT.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus type: chronic, subjective, non - pulsatile tinnitus
* Duration of tinnitus = more than 3 months
* Minimum age of the patient is 18 years old - maximum age is 75 years old
* Tinnitus Functional Index (TFI) score ≥ 25 - < 90
* Stable use of medication during therapy

Exclusion Criteria:

* HADS - score: anxiety and depression-subscores > 15
* HQ - score > 40
* Objective, pulsatile tinnitus
* Active middle ear pathology
* Neurological and psychiatry co-morbidity for which currently psychotherapy is ongoing
* Psychosis, schizophrenia, epilepsy
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-10; Primary Completion 2019-09 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) | Change will be assessed at 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2). The change will be assessed at every test moment.
  The TFI is a self-reported questionnaire, consisting of 25 questions, which assesses the impact of tinnitus on patients' daily lives. The patient answers each question on a Likert scale ranging from 0 to 10. Questions 1 and 3 are expressed in percentages, and the Likert scale ranges from 0 % to 100 %. The total score is calculated with the mean of all questions. The answers are converted and the total score is expressed as a number between 0 and 100. In addition to the total score, the score of eight subscales can be determined. The subscales are the following: intrusiveness, reduced sense of control, cognitive interference, sleep disturbance, auditory difficulties attributed to tinnitus, interference with relaxation, reduced quality of life and emotional distress.
  A decrease in the score on the TFI in the TRT-CBT-treatment group versus a decrease in the TFI-score in the TRT- EMDR-treatment group is the primary focus of attention in this study.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of loudness | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).The secondary outcome measurements will be assessed at every test moment.
  The patient scores the mean and maximum loudness of their tinnitus on a scale of 0 (absence of tinnitus) to 10 (as loud as possible, cannot be any louder).
Tinnitus questionnaire (TQ) | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).The secondary outcome measurements will be assessed at every test moment.
  The TQ is a 52-item self-rating scale, which differentiates between dimensions of emotional and cognitive distress, intrusiveness, auditory perceptual difficulties, sleep disturbances and somatic complaints. The patient rates the items on a 3-point scale.
Hospital Anxiety and Depression Scale (HADS) | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).The secondary outcome measurements will be assessed at every test moment.
  The HADS consists of 14 questions that assess anxiety and depression. The patient can choose between four answer options for each question. The score for both components is a summation of the scores of all the questions belonging to the subscale. A result greater than 8 suggests the presence of a depression and/or anxiety disorder.
Hyperacusis Questionnaire (HQ) | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).The secondary outcome measurements will be assessed at every test moment.
  The HQ is a 14-item questionnaire that surveys a patient's hypersensitivity to sound. There are four answer options for every question: 'no', 'yes a little', 'yes quite a lot' and 'yes a lot'. A score of 28 is the cut-off for auditory hypersensitivity.
Psychoacoustic measurements | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).These measurements will only be used to evaluate within-patient variability.
  In order to categorize our patient group, all subjects will undergo an audiometric hearing test according to current clinical standards (International Organisation for Standardization (ISO) 8253-1:2010) with a 2-channel Interacoustics AC 40 (Interacoustics A/S, Middelfart, Denmark) in a soundproof audiometric booth. The TDH-39 headphone is used as transducer to measure air conduction thresholds of frequencies ranging from 125 Hz to 8 kHz. If air conduction thresholds exceed 20 dB HL, bone conduction thresholds will be determined within a range of 250 Hz to 4 kHz.
  The frequency of tinnitus will be determined by means of frequency matching for which a forced choice technique is applied. The patient must choose between two presented tones or noises until a tone or noise is found that is similar to the patient's tinnitus.
ERP | There will be 3 test moments during the trial: before the start of therapy (T0), after 3 months (10 treatment sessions) (T1) and 3 months after the last therapy session (T2).The secondary outcome measurements will be assessed at every test moment.
  In this study, the emphasis is on the late auditory evoked potentials which will be evoked by use of a classical oddball paradigm. As such a standard tone of 1 kHz is repeated with a probability of 80% randomly interrupted by an oddball (or infrequent) tone of 2 kHz with a probability of 20%. This paradigm elicits late auditory evoked potentials comprising of P1-N1-P2 and P300 of which the first complex is mostly generated by bottom-up processes in the brain. The later P300 potential requires more top-down cognitive brain processes and can be seen as an expression of higher cognitive sound processing in tinnitus patients. The hypothesis is that, given the continuous auditory processing of the tinnitus signal, the brain may have less capacity left to align to other incoming stimuli which may be altered by therapy.
  The late auditory potentials will be measured prior to the therapy, after the therapy and 3 months later.
Big Five Inventory - 2 (BFI) | Timeframe within 12 months
  BFI-2 (Soto & John, 2017) is self-report questionnaire contains 60 items with a forced-choice of 5 items (e.g. totally disagree - disagree - don't agree/don't disagree - agree - totally agree).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Paul Van de Heyning, MD PhD, Study Director — Chairman dept of ENT and Head and Neck Surgery, Antwerp University Hospital
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Luyten TR, Jacquemin L, Van Looveren N, Declau F, Fransen E, Cardon E, De Bodt M, Topsakal V, Van de Heyning P, Van Rompaey V, Gilles A. Bimodal Therapy for Chronic Subjective Tinnitus: A Randomized Controlled Trial of EMDR and TRT Versus CBT and TRT. Front Psychol. 2020 Sep 10;11:2048. doi: 10.3389/fpsyg.2020.02048. eCollection 2020. PMID 33013517
- [Derived] Luyten T, Van de Heyning P, Jacquemin L, Van Looveren N, Declau F, Fransen E, Gilles A. The value of Eye Movement Desensitization Reprocessing in the treatment of tinnitus: study protocol for a randomized controlled trial. Trials. 2019 Jan 9;20(1):32. doi: 10.1186/s13063-018-3121-6. PMID 30626414